CLINICAL TRIAL: NCT02172105
Title: A Double-blind, Randomised, Placebo Controlled (Within a Dose Group) Study to Evaluate Safety, Tolerability and Pharmacokinetics of Multiple Rising Inhalative Doses (5 μg, 10 μg and 20 μg) of BI 1744 CL for 14 Days in Healthy Male Volunteers
Brief Title: Multiple Rising Inhalative Doses of BI 1744 CL in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.21
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol

ARMS (2):
- BI 1744 CL (Experimental)
  Interventions: Drug: BI 1744 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: BI 1744 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate safety, tolerability, and pharmacokinetics of BI 1744 CL in healthy Japanese male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese men: According to the results of a complete medical history, the physical examination, vital signs (blood pressure and pulse rate), 12-lead ECG, clinical laboratory tests
* Age ≥20 and ≤35 years
* Body mass index (BMI) ≥18.5 and ≤25.0 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation
* Subjects must be able to inhale medication in a competent manner from the Respimat®inhaler

Exclusion Criteria:

* Any finding of the medical examination (including ,blood pressure and pulse rate and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug before drug administration or during the trial
* Use of prescription or non-prescription drugs within 10 days before drug administration or during the trial. However, over-the-counter drugs for external application (such as lubricant eye drops for contact lens, insect bite reliever) shall be allowed
* Participation in another trial with an investigational drug within four months before drug administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day: corresponds to ca. 3 large bottles of beer, 3 gous (ca. 540 cc) of Japanese sake, 6 shots of whisky, 6 glasses of wine or 6 glasses of Japanese shochu, distilled alcoholic beverage)
* Drug abuse
* Blood donation (more than 100 mL within four weeks before drug administration or during the trial)
* Excessive physical activities (within one week before administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms) or long QT syndroms
* A history of additional risk factors for torsades de pointes (TdP) (e.g., heart failure, hypokalemia) or other cardiac arrhythmias
* hyperthyroidism
* Disagree with adequate contraception (the subject should use condoms and his partner should use oral contraception or intrauterine device [IUD]) during the study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline, up to 13 days after last drug administration
Number of patients with clinically relevant findings in vital signs (blood pressure, pulse rate) | Baseline, up to 13 days after last drug administration
Number of patients with abnormal findings in 12-lead electrocardiogram (ECG) | Baseline, up to 13 days after last drug administration
Number of patients with clinically significant changes in clinical laboratory tests | Baseline, up to 13 days after last drug administration
Change from baseline in potassium level | Baseline and Day 14
Number of patients with adverse events | 7 weeks
Assessment of tolerability on a 4-point scale | Day 28

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma at different time points) | Up to day 18
tmax (time from dosing to maximum measured concentration of the analyte in plasma at different time points) | Up to day 18
AUC (area under the concentration-time curve of the analyte in plasma at different time points) | Up to day 18
%AUCtz-∞ (the percentage of the AUC 0-infinity that is obtained by extrapolation) | Up to day 18
λz (terminal rate constant in plasma at different time points) | Up to day 18
t1/2 (terminal half-life of the analyte in plasma at different time points) | Up to day 18
MRTih (mean residence time of the analyte in the body after inhalation administration at different time points) | Up to day 18
Aeτ (amount of analyte that is eliminated in urine after administration over a uniform dosing interval τ at different time points) | Up to day 18
feτ (fraction of analyte eliminated in urine after administration over a uniform dosing interval τ at different time points) | Up to day 18
CLR (renal clearance of the analyte at different time points) | Up to day 18
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to day 18
Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | Up to day 18
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to day 18
CL/F,ss (apparent clearance of the analyte in the plasma at steady state following extravascular multiple dose administration) | Up to day 18
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | Up to day 18
Accumulation ratio (RA,AUC) | Up to day 18
Accumulation ratio (RA,Cmax) | Up to day 18